CLINICAL TRIAL: NCT04197466
Title: Comparison of Different Treatments for Overactive Bladder Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/06/09
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Overactive Detrusor
Keywords: Pelvic Floor Muscle Exercise; Kinesio taping; Electric Stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Athletic Tape; Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pelvic Floor Exercise Group (Experimental): Pelvic floor muscle exercises will be recommended as a home program for 6 weeks every day of the week.
  Interventions: Other: Pelvic Floor Exercise Group
- Kinesiotape Group (Experimental): In addition to pelvic floor exercise,kinesio tape application will be performed by ligament technique to the sacral region.
  Interventions: Other: Pelvic Floor Exercise Group; Other: Kinesio tape
- Electrical Stimulation Group (Experimental): In addition to pelvic floor exercise,electrical stimulation will be performed in the lying, sitting, stand up positions for 30 minutes
  Interventions: Other: Pelvic Floor Exercise Group; Other: Electrical stimulation

INTERVENTIONS:
Other: Pelvic Floor Exercise Group — The exercise program will be tailored according to the pelvic floor muscle strength, including fast and slow contractions. The number and duration of exercises will be increased according to progress..
Other: Kinesio tape — Kinesio tape application will be performed by ligament technique to the sacral region.
  Arms: Kinesiotape Group
Other: Electrical stimulation — External electrical stimulation will be performed in the lying, sitting, stand up positions for 30 minutes
  Arms: Electrical Stimulation Group

SUMMARY:
This study aims to investigate the effects of pelvic floor muscle exercises, electrical stimulation and taping in patients with overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Women
* Being Volunteered to participate
* Diagnosed as overactive bladder

Exclusion Criteria:

* Pregnant women
* Patients with a comorbid neurological disorder
* A mental problem that may prevent cooperation and evaluation
* Acute infection
* Sensory loss
* Malignancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Bladder Diary | Before the treatment, at end of 6 weeks
  Women will be asked to complete a 24-hour frequency-volume chart (urine diary) to assess bladder symptoms. Each woman will fill the chart for a total of 3 days filled in 3 consecutive days. In these diaries, women will be asked to record the number of their urination during the day, how much urine they produce each time they urinate, their incontinence, the type and amount of drinks. Women will be warned not to change their daily voiding habits and the amount of fluids they consume during filling these charts. The data obtained from these three days will be averaged to determine daily voiding frequency, night voiding frequency, average voiding volume, and daily urinary incontinence.

SECONDARY OUTCOMES:
King Health Questionnaire | Before the treatment and end of 6 weeks
  The Turkish version of the King Health Questionnaire, which was developed to assess the quality of life of women, consisting of 21 items, was shown to be valid and reliable The survey consists of 3 sections and 9 sub-headings. These subheadings are questions that determine general health perception, incontinence impact, role, physical and social limitations, personal relationships, emotions, sleep / energy and severity measures. In addition, the third section includes 9 questions that question the effect of urinary symptoms. In each subheading, a complex scoring algorithm is used for missing values. Scoring varies between "0" and "100.. Decrease in score indicates an increase in quality of life
Pelvic Floor Muscle Strength | Before the treatment and end of 6 weeks
  Modified Ashword Scale and perineometer device will be used for the measurement of the pelvic floor muscle strength. Modified Ashword Scale is a 6-point scale: 0=no contraction, 1=flicker, 2=weak, 3=moderate, 4=good (with lift), and 5=strong. This measurement scale is incorporated with vaginal palpation in the clinical assessment,.
  The PFX perineometer (Cardio Design Pty Ltd, Australia) will be used to provide an objective measurement. In the lithotomy position the probe of the perineometer will be inserted into the vagina of the patient. The patient will be asked to relax and squeeze the probe of the perineometer as if they are holding the urine or gaita. The minimum and maximum value of the perineometer are between 0-12 kg Pascal (kPa) and the difference between the first value and the last value in the perineometer will be determined as the pelvic floor muscle strength. The average of three repetitions will be noted
Overactive bladder symptoms | Before the treatment, at end of 6 weeks
  Symptoms will be assessed by the Turkish version of the Overactive Bladder-V8 (OAB-V8) questionnaire, which has been shown to be valid and reliable. The AAM-V8 questionnaire had 8 questions scored as 0 to 5. The total score ranges from 0 to 40. Increased scores indicate that the severity of overactive bladder complaints increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt Üniversitesi, Ankara, Turkey (Türkiye)